CLINICAL TRIAL: NCT03494764
Title: Hyperbaric Oxygen Therapy for Moderate to Severe Ulcerative Colitis Flares: A Multi-Center Randomized Trial
Brief Title: Hyperbaric Oxygen Therapy for Ulcerative Colitis Flares
Acronym: HBO-UC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Foundation for Clinical Research in IBD (Unknown); The Eli and Edythe Broad Foundation (Unknown); University of California, San Diego (Other); Mayo Clinic (Other); University of Pittsburgh Medical Center (Other); Virginia Mason Memorial Hospital (Unknown); University of Texas Southwestern Medical Center (Other); University of Maryland, College Park (Other); NYU Langone Health (Other)
Responsible Party: Principal Investigator, Corey Siegel, Section Chief, Section of Gastroenterology, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Broad-IBD-HBO-UC D12161
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Colitis, Ulcerative
Keywords: Hyperbaric Oxygen Therapy
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 Days Hyperbaric Therapy (Active Comparator): Patients will be enrolled and follow an identical medical treatment algorithm. At day 3 responders (based on partial Mayo score) will be re-randomized in a 1:1 fashion to complete 5 total days of HBOT (1 session per day) or to stop after 3 days of HBOT. Non-responders will be entered into an open label arm to complete 5 total days of HBOT.
  Interventions: Other: Hyperbaric Oxygen Therapy
- 3 Days Hyperbaric Therapy (Active Comparator): Patients will be enrolled and follow an identical medical treatment algorithm. At day 3 responders (based on partial Mayo score) will be re-randomized in a 1:1 fashion to complete 5 total days of HBOT (1 session per day) or to stop after 3 days of HBOT. Non-responders will be entered into an open label arm to complete 5 total days of HBOT.
  Interventions: Other: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Other: Hyperbaric Oxygen Therapy — Hyperbaric oxygen (HBO) provides 100% oxygen at a pressure above atmospheric pressure (typically twice to three times standard sea level pressure (2.0-3.0 ATA)). This dramatically increases the amount of oxygen dissolved in blood plasma, which in turn increases oxygen delivery to tissues. This effect of hyperbaric oxygen is used clinically to treat acute hypoxia in crush injuries, severed limbs, and failing skin grafts

SUMMARY:
Ulcerative colitis (UC) is a chronic inflammatory bowel disease associated with recurrent mucosal inflammation. Clinically, the disease is characterized by bloody diarrhea, abdominal pain, and constitutional symptoms such as fever and weight loss. Treatment strategies vary based on disease activity and target various aspects of the inflammatory cascade. Options include: anti-inflammatory drugs (mesalamine), immunosuppressive or modulatory medications (corticosteroids, thiopurines, cyclosporine) and biologic agents (Anti-TNF). Disease severity can be wide ranging, and nearly 25% of UC patients are hospitalized for acute severe disease. Of these patients, 30% will undergo colectomy after the acute episode, a quarter of which will experience post-operative complications. Although there has been great progress in treatment of UC over the past decade, even with the anti-TNF agent infliximab, the one-year remission rate for patients not responding to conservative management is barely 20%. Furthermore, corticosteroids have significant long-term consequences and immune suppressive drugs such as 6-mercaptopurine, azathioprine and infliximab have been associated with serious adverse events including life-threatening infections and lymphomas. With growing evidence that the pathogenesis of UC is multi-factorial and involves a complex interaction of genetic and environmental factors, newer treatment modalities are being evaluated to target the mucosal immune response and mucosal inflammatory regulatory system.

Hyperbaric oxygen offers a promising new treatment option since it targets both tissue hypoxia and inflammation. Recent small scales studies evaluating the impact of hyperbaric oxygen treatment in acute ulcerative colitis flares demonstrated improved outcomes. The mechanisms underlying the improvement are not known. In this study, we will treat ulcerative colitis flares with hyperbaric oxygen and measure changes in both markers of tissue hypoxia and inflammation. We hypothesize that hyperbaric oxygen will (a) improve outcomes, and (b) show reductions in markers of both tissue hypoxia and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with known or newly diagnosed moderate to severe ulcerative colitis (as defined by the Mayo score ≥6)
* Consented within the first 48 hours of initiating IV steroids
* Risk score of >3 points (pts)

  * Mean stool frequency/24 hrs (<4 = 0 pts, 4-6 = 1 pt, 7-9 = 2 pts, >9 = 4 pts)
  * Colonic Dilation = 4pts
  * Hypoalbuminemia (< 3mg/dL) = 1 pts
* Mayo endoscopic sub-score >2 (moderate to severe)
* Age >18 and able to make their own medical decisions

Exclusion Criteria:

* Complication requiring urgent surgical intervention (in the opinion of the investigators)
* Clinically significant cardiac, renal, neurological, endocrine, respiratory or hepatic impairment in the opinion of the investigator, including but not limited to:

  * Pulmonary (COPD with CO2 retention; Previous/current imaging showing hyperinflation/air trapping/bullous disease/blebs (opinion of investigators), Current pneumothorax or previous spontaneous pneumothorax, Bronchogenic cyst(s))
  * Cardiac (Uncontrolled HTN (systolic >160 or diastolic >100), Unstable angina or myocardial infarction within the previous 3 months, Ejection fraction < 35%, Current or previous amiodarone use, ICD in place, Pacemaker in place not approved for chamber use)
  * Hematological/Oncological (Current chemotherapeutic drug use, and past history of bleomycin use,Hereditary Spherocytosis, Sickle cell anemia)
  * Gastrointestinal and Infectious Disease (Known or suspected Crohn's disease, Previous infection with mycobacterium, fungus, HIV, Hepatitis B or C, Severe gastrointestinal or systemic infection (opinion of investigator), Current capsule endoscopy or previously non-retrieved capsule
  * Endocrinology (Uncontrolled hyperthyroidism)
  * Neurological and Psychological (Vagal or other nerve stimulators, Uncontrolled seizure disorder, Medications or medical conditions that lower seizure threshold (opinion of the investigator), Drug or alcohol abuse/dependence,Current treatment for alcohol cessation with disulfiram, Current or recent (within past week) use of baclofen)
  * Head and Neck (Previous middle ear damage, surgery or infection(s) which may increase the risk for needing ear tubes (opinion of the investigator),Current or previous retinal detachment or optic neuritis, Retinal or vitreous surgery within the past 3 months)
* Implanted devices not on the approved list for use with HBOT
* Women who are pregnant or nursing. Women with childbearing potential were required to use effective birth control if not surgically sterile or postmenopausal for >2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Impact of HBOT on clinical response/remission | 5 Days
  Impact of HBOT on clinical response/remission to medical therapy as measured by the partial Mayo score at study day 5.

SECONDARY OUTCOMES:
relative and absolute reduction in the Mayo score | Day 5, 10
  Relative and absolute reduction in the Mayo score
Flair duration | day 5, 10
  time to reduction in mayo score
Hospitalization duration | day5, 10
  time in the hospital
proportion of patients requiring other therapy | Day 5, 10
  Proportion who require cyclosporine, infliximab or colectomy during index flare
Relative and absolute change in inflammatory markers | day 10
  Relative absolute change in inflammatory markers: ESR
Relative and absolute change in inflammatory markers | day 10
  Relative absolute change in inflammatory markers: CRP
Relative and absolute change in inflammatory markers | day 10
  Relative absolute change in inflammatory markers: fecal calprotectin
Relative and absolute change in inflammatory markers | day 10
  Relative absolute change in inflammatory markers: interleukins
Relative and absolute change in gene expression | day 10
  Relative absolute change in gene expression: VEGF
Relative and absolute change in gene expression | day 10
  Relative absolute change in gene expression: HIF-1
Relative and absolute change in gene expression | day 10
  Relative absolute change in gene expression: HO-1
microbiome composition | day 10
  Describe the HBOT specific changes in the microbiome composition

CONTACTS AND LOCATIONS:
Overall Officials: Parambir Dulai, MD, Principal Investigator — University of California, San Diego
Locations (8):
- United States (8):
  - UC San Diego Health Systems, La Jolla, California
  - University of California San Diego, San Diego, California
  - University of Maryland, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Langone Medical Center, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Virginia Mason Memorial Hospital, Yakima, Washington